CLINICAL TRIAL: NCT01319578
Title: A Single Blind Pharmacodynamic Study to Assess the Phosphate Binding Characteristics of K2CG Chewing Gum
Brief Title: PD Study to Assess Phosphate Binding Characteristics of K2CG Chewing Gum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Nephrologists, P.C. (Other)
Collaborators: CM&D Pharma Limited (Industry)
Responsible Party: Geoffrey A. Block, MD, Principal Investigator, Denver Nephrologists, PC
Allocation: Non-Randomized | Model: Crossover | Masking: Single
Other Study IDs: CMD 005
Record Dates: First submitted 2011-03-03; First posted 2011-03-21 (Estimated); Last update posted 2011-11-15 (Estimated); Status verified 2011-11

CONDITIONS: Hyperphosphatemia; Chronic Kidney Disease
Keywords: chronic kidney disease; phosphorus; phosphate; saliva; K2CG; medical food; chitosan
MeSH Terms: conditions — Hyperphosphatemia; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Chewing Arm 1 (Active Comparator)
  Interventions: Other: K2CG chewing gum
- Chewing Arm 2 (Placebo Comparator)
  Interventions: Other: K2CG chewing gum
- Chewing Arm 3 (Active Comparator)
  Interventions: Other: K2CG chewing gum
- Chewing Arm 4 (Active Comparator)
  Interventions: Other: K2CG chewing gum

INTERVENTIONS:
Other: K2CG chewing gum — Fasting: Chew gum 15 minutes Post meal: Begin chewing 45 minutes post meal
Other: K2CG chewing gum — Fasting: Chew gum 30 minutes Post meal: Begin chewing 30 minutes post meal
Other: K2CG chewing gum — Fasting: Chew gum for 45 minutes Post meal: Begin chewing gum 15 minutes post meal
Other: K2CG chewing gum — Fasting: Chew gum for 60 minutes Post meal: Being chewing gum 5 minutes post meal

SUMMARY:
The specific purpose of this study is to describe the characteristics of the K2CG chewing gum, specifically as it relates to duration of gum chewing (exposure), timing of gum chewing in relation to a meal, and dose of K2CG chewing gum.

DETAILED DESCRIPTION:
Previous studies have demonstrated that salivary phosphate levels are elevated in patients with CKD and that there is a direct and linear correlation between serum phosphorus and salivary phosphorus. K2CG chewing gum may provide an alternative approach to treating patients with elevated phosphate levels. However, data regarding the pharmacodynamic effect of the K2CG chewing gum on salivary phosphorus is lacking; as such, this study seeks to examine the phosphate binding characteristics of K2CG chewing gum with 2 different amounts of chitosan and varying exposure time in the fasting and fed condition.

A precise knowledge of the pharmacodynamic effect of the K2CG chewing gum on salivary phosphorus is expected to provide information necessary to plan and conduct a subsequent interventional trial with K2CG chewing gum in patients with both Chronic Kidney Disease and ESRD. Specifically, quantification of the amount of salivary phosphorus that binds to 3 formulations of chitosan loaded chewing gum (20 mg, 40 mg and 60 mg) with varying exposure times will inform the optimal duration of exposure relative to gum size. The effect of gum size will be further explored via the use of two different sizes of placebo chewing gum (1.7 g and 2.0 g sizes). Additionally it is a specific aim of this study to assess whether chewing gum in the fasted vs. fed state affects the binding characteristics of chitosan loaded chewing gum.

This study is a pharmacodynamic study to characterize the phosphate binding capabilities of three different doses of K2CG chewing gum (20mg, 40mg, 60mg) and one placebo chewing gum (1.7 g). Thirty-six subjects will be enrolled across three renal function group based on estimated glomerular filtration rate.

Study assessments will occur over four study visit days (Visit 2, Visit 3, Visit 4, and Visit 5). Fasting study procedures will occur in the morning of each visit day, and non-fasting procedures will occur following the administration of a standardized meal on the same day. All subjects will receive three doses of K2CG chewing gum and one placebo: 20 mg dose at Visit 2, 1.7 g placebo at Visit 3, 40 mg dose at Visit 4, and 60 mg dose at Visit 5. Subjects will not be aware of the specific gum dose or size at any study visit (single blind). The duration of gum chewing and timing of salivary collections will vary within each group.

Saliva will be collected at specified time points throughout the trial. Fasting salivary phosphorus must be collected with nothing to eat or drink for at least 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Men or women > 18 years of age;
* Must have no dietary restriction that would preclude eating standardized meal (both a meat based and vegan option available)
* The subject has voluntarily signed and dated the most recent informed consent form approved by an Institutional Review Board (IRB).
* Must be able to chew gum for at least 60 minutes.
* Must have historical eGFR appropriate for the study.

Exclusion Criteria:

* Receiving or has received an investigational product (or is currently using an investigational device) within 30 days prior to Visit 2;
* Evidence of active (clinically significant) infection at the time of study enrollment (in the opinion of the investigator);
* Dental work within 48 hours of enrollment (Visit 2); and
* Known sensitivity to chitin, or allergy to shellfish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
total phosphate bound per gum piece fasting | 15 min, 30 min, 45 min, 60 min post chewing
  patients will be assigned to treatment arms of varying chewing duration fasting and the total phosphorous bound per piece of chewing gum will be assessed. each patient will recieve (in random order) gum with placebo, 20 mg, 40 mg, and 60 mg chitosan content
total phosphate bound per piece of gum post meal | 5 min, 15 min, 30 min, 45 minutes post meal
  Each subject will begin chewing at the assigned time post meal exposure and chew for 30 minutes. total phosphorus bound per piece of gum will be assessed. each patient will recieve (in random order) gum with placebo, 20 mg, 40 mg, and 60 mg chitosan content

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey A Block, MD, Principal Investigator — Denver Nephrologists, PC
Locations (1):
- Denver Nephrologists, PC, Denver, Colorado, United States

REFERENCES:
- [Derived] Block GA, Persky MS, Shamblin BM, Baltazar MF, Singh B, Sharma A, Pergola P, Smits G, Comelli MC. Effect of salivary phosphate-binding chewing gum on serum phosphate in chronic kidney disease. Nephron Clin Pract. 2013;123(1-2):93-101. doi: 10.1159/000351850. Epub 2013 Jun 22. PMID 23797006